CLINICAL TRIAL: NCT00752908
Title: Tissue Penetration of Antibiotics in Obesity
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 070678
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, interstitial fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese patients: Obese patients
- Normal weight patients and volunteers: Normal weight patients and volunteers

SUMMARY:
The purpose of this study is to evaluate cefoxitin pharmacokinetics in obese surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI <25 and >40
* Scheduled for elective abdominal or pelvic surgery
* Surgical plan for intraoperative cefoxitin prophylaxis
* Able to provide informed consent

Exclusion Criteria:

* Allergy to Cefoxitin
* Renal or Hepatic insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical Patients at BJH
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan D Kharasch, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obese Patients | Normal Weight Patients and Volunteers
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Patients | Normal Weight Patients and Volunteers | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 28 (12) | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 2 | 6 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Cefoxitin Plasma Concentrations
Description: Cefoxitin plasma concentrations
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: (µg/mL)
Arm/Group | Obese Patients | Normal Weight Patients and Volunteers
Number analyzed (Participants) | 14 | 13
(µg/mL) | 89 (20) | 81 (33)
Statistical Analysis 1: Comparison: Obese Patients vs Normal Weight Patients and Volunteers; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Cefoxitin Tissue Concentrations
Description: Cefoxitin tissue concentrations
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: (µg/mL)
Arm/Group | Obese Patients | Normal Weight Patients and Volunteers
Number analyzed (Participants) | 10 | 10
(µg/mL) | 8.8 (6.6) | 26 (20)

ADVERSE EVENTS:
Arm/Group | Obese Patients | Normal Weight Patients and Volunteers
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes